CLINICAL TRIAL: NCT02451865
Title: A Phase IB Dose Escalation and Expansion Trial of MEK 162 With Docetaxel in Previously Treated Stage IV, Non-small Cell Lung Cancer (NSCLC)
Brief Title: Binimetinib With Docetaxel in Treating Patients With Previously Treated, Stage IV Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-001595; NCI-2015-00618 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Garon MEK162 NSCLC (Other: Jonsson Comprehensive Cancer Center); 14-001595 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2016-07

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — binimetinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (binimetinib and docetaxel) (Experimental): Patients receive binimetinib PO BID on days 1-21 and docetaxel IV on day 21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who have stable disease or better after completing 6 courses of binimetinib and docetaxel may continue receiving binimetinib PO BID in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Drug: Docetaxel; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162
Drug: Docetaxel — Given IV
  Other Names: RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase Ib trial studies the safety and best dose of binimetinib when given in combination with docetaxel in treating patients with previously treated, stage IV non-small cell lung cancer. Binimetinib and docetaxel may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of increasing doses of MEK162 (binimetinib) with docetaxel 75 mg/m2 every 21 days in patients with stage IV non-small cell lung cancer (NSCLC) that have progressed after at least one prior systemic therapy.

SECONDARY OBJECTIVES:

I. Determine objective tumor response rate (RR) as defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 with MEK162 and standard doses of docetaxel in stage IV NSCLC.

II. Determine progression free survival (PFS) of MEK162 and standard doses of docetaxel.

III. Evaluate the pharmacokinetic profile of MEK162 when given along with docetaxel.

TERTIARY OBJECTIVES:

I. Evaluate tissue biomarkers in baseline tumors and at the time of progression to correlate with clinical outcome II. Assess the activation status of extracellular signal-regulated kinase (ERK), protein kinase B (Akt) and ribosomal protein S6 kinase (S6K) in tumor biopsy samples at baseline and at the time of progression.

III. Determine the cytokine profile before and after treatment in patients.

OUTLINE: This is a dose-escalation study of binimetinib.

Patients receive binimetinib orally (PO) twice daily (BID) on days 1-21 and docetaxel intravenously (IV) on day 21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who have stable disease or better after completing 6 courses of binimetinib and docetaxel may continue receiving binimetinib PO BID in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* A histologically or cytologically confirmed diagnosis of stage IV NSCLC
* Must have progressed on at least one prior line of platinum-based therapy for stage IV NSCLC (excluding docetaxel or mitogen activated protein kinase kinase [MEK] inhibitors)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Measurable disease defined by RECIST criteria
* Ability to provide adequate tissue from archival tumor specimen; confirmation of adequate tissue is required prior to enrollment
* In expansion cohort only: patient's kirsten rat sarcoma viral oncogene homolog (KRAS) mutational status must be known prior to enrollment
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin (Hgb) >= 9 g/dL without transfusions
* Platelets (PLT) >= 100 x 10^9/L without transfusions
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 1.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN
* Creatinine =< 1.5 mg/dL
* Left ventricular ejection fraction (LVEF) >= 45% as determined by a multigated acquisition (MUGA) scan or echocardiogram, and QTc interval =< 480ms
* Able to take and retain oral medications
* Patient is deemed by the investigator to have the initiative and means to be compliant with the protocol (treatment and follow-up)
* Negative serum beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only) performed locally within 72 hours (hrs) prior to first dose

Exclusion Criteria:

* History or current evidence of retinal vein occlusion (RVO) or current risk factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
* History of Gilbert syndrome
* Previous or concurrent malignancy within the last 3 years with the exception of adequately treated skin basal or squamous cell with adequate wound healing
* Prior therapy with a MEK-inhibitor or docetaxel for metastatic non-small cell lung cancer (docetaxel in the adjuvant setting will be allowed)
* Epidermal growth factor receptor (EGFR) mutant and/or anaplastic lymphoma receptor tyrosine kinase (ALK) gene rearranged tumor
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following within 6 months of enrollment: myocardial infarction, unstable angina, coronary artery bypass graft (CABG), coronary angioplasty, or stenting, symptomatic chronic heart failure, clinically significant cardiac arrhythmias and/or conduction (except atrial fibrillation and paroxysmal supraventricular tachycardia)
* Uncontrolled arterial hypertension despite appropriate medical therapy
* Known positive serology for human immunodeficiency virus (HIV), active hepatitis B, and/or active hepatitis C infection
* Neuromuscular disorders that are associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy)
* Subjects planning on embarking on a new strenuous exercise regimen after first dose of study treatment that can result in significant increases in plasma CK levels
* Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption)
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to concerns regarding safety or compliance with clinical study procedures
* Patients who have undergone major surgery =< 3 weeks prior to starting study drug or who have not recovered from side effects of such procedure
* Pregnant or lactating women
* Women of child-bearing potential defined as all women physiologically capable of becoming pregnant who are unwilling to use highly effective methods of contraception throughout the study and 15 days after study drug discontinuation
* Sexually active males unless they are willing to use a condom during intercourse while taking the drug and for 15 days after stopping treatment and are willing to forego fathering a child in this period; a condom is required to be used also by vasectomized men
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study
* Grade II or greater neuropathy at baseline
* Symptomatic brain metastases (if a patient has brain metastases and is on steroids, the steroid dose must have been stable for at least 14 days) or brain metastases that have not been previously treated
* Treatment with prior chemotherapy, monoclonal antibodies, other protein or peptide therapeutics or anticancer immunotherapy within 21 days of the first dose of study drug
* Treatment with prior radiotherapy within 28 days of initiating study drug; however, if the radiation portal covered =< 10% of the bone marrow reserve, the patient may be enrolled without respect to the end date of radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03 | Up to 30 days post-treatment
  Side effects will be tabulated according to grade and will do sub-analysis based on patient demographic categories such as age and ECOG performance status.
Incidence of dose-limiting toxicities, graded according to the CTCAE v4.03 | 21 days
  Side effects will be tabulated according to grade and will do sub-analysis based on patient demographic categories such as age and ECOG performance status.
Maximum tolerated dose of binimetinib in combination with docetaxel | 21 days

SECONDARY OUTCOMES:
Biomarker analyses | Up to 30 days post-treatment
  Will determine if there is a correlation of baseline biomarkers and objective tumor response. For categorical markers will use Fisher's exact test to examine the relationship with response and different categorical variables at specific time points. For quantitative markers will use one-way analysis of variance to compare the marker levels between response categories. Correlations between pairs of quantitative markers will be performed using Pearson correlations if the marker distributions are approximately normal. For non-normality will use the Kendall correlation coefficients.
Mutations in KRAS and NRAS | Up to 30 days post-treatment
  Will determine if there is a correlation of response in patients treated with docetaxel and binimetinib with mutations in KRAS and NRAS.
Objective tumor response rate (the rate of complete response or partial response), as defined by RECIST 1.1 | Up to 5 years
  The proportion ever achieving a clinical and objective tumor response will be estimated and will construct an exact one-sided 90% confidence interval to identify the likely range for the underlying tumor response rate. Tumor response will be correlated with biomarkers as well as other patient characteristics such as ECOG performance status, k-ras and neuroblastoma RAS viral oncogene homolog (n-ras) mutational status using a variety of analytic techniques.
Pharmacokinetic (PK) profile will assess binimetinib (MEK162) levels during treatment cycles | On days 1 and 8 of course 1 and on day 1 of course 2
  Analyzed by tabulation of PK values with mean and standard deviation at each time point.
Progression free survival | Up to 5 years
  Cox-proportional hazards regression models will be used to correlate time to disease progression to both quantitative and categorical variables. Survival distributions will be estimated with the Kaplan-Meier method and significant differences between survival rates will be calculated with the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garon, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States